CLINICAL TRIAL: NCT05329272
Title: Effects of Incorporating Virtual Reality Training Intervention Into Health Care on Cognitive Function and Quality of Life in Older Adults With Cognitive Impairment: A Randomized Controlled Trial
Brief Title: Virtual Reality Training Intervention on Cognitive Function and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I-Shou University (Other)
Responsible Party: Principal Investigator, Mei-Chi Hsu, Professor, I-Shou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IShouU-VR
Record Dates: First submitted 2022-03-21; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Virtual Reality; Cognitive Impairment; Quality of Life
Keywords: Virtual Reality; Cognitive Impairment; Quality of Life; Long-term care facilities
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The VR group: the Virtual Reality Cognitive Training Intervention (VRCTI) (Experimental): The VRCTI was developed to improve cognitive function. The intervention was designed that simulated schema of underwater world fish swimming. Each 1-hour session was typically divided into three parts: easy, medium and difficult, each with 4 different tasks, so there are 12 tasks/session in total. In some tasks, the VRCTI also distinguished between the real lure (e.g. a red triangle fish with a half-moon pattern) as well as unrelated lure items (i.e., blue square fish with polka dot pattern and other irrelevant items). The use of hardware elements for this study included visual (head-mounted display [HMD] in delivering the VR intervention), audio, and motor equipment.
  Interventions: Other: Virtual Reality Cognitive Training Intervention (VRCTI)
- The control group (No Intervention): The control group received usual care.

INTERVENTIONS:
Other: Virtual Reality Cognitive Training Intervention (VRCTI) — The VRCTI was developed to improve cognitive function. The intervention was designed that simulated schema of underwater world fish swimming. Each 1-hour session was typically divided into three parts: easy, medium and difficult, each with 4 different tasks, so there are 12 tasks/session in total. In some tasks, the VRCTI also distinguished between the real lure (e.g. a red triangle fish with a half-moon pattern) as well as unrelated lure items (i.e., blue square fish with polka dot pattern and other irrelevant items). The use of hardware elements for this study included visual (head-mounted display [HMD] in delivering the VR intervention), audio, and motor equipment.
  Arms: The VR group: the Virtual Reality Cognitive Training Intervention (VRCTI)

SUMMARY:
The present study aimed to investigate the effects of a Virtual Reality cognitive training intervention (VRCTI) on cognitive function changes measured with a cognitive test battery and improvement of quality of life in older adults with cognitive impairment in long-term care facilities. Weekly 1-hour sessions were implemented over 8 weeks targeting sustained and selective attention, memory, cognitive functions, and rule deduction. The passive control group received usual care.

DETAILED DESCRIPTION:
Objectives: The present study aimed to investigate the effects of a Virtual Reality cognitive training intervention (VRCTI) on cognitive function changes measured with a cognitive test battery and improvement of quality of life in older adults with cognitive impairment in long-term care facilities.

Method: Weekly 1-hour sessions were implemented over 8 weeks targeting sustained and selective attention, memory, cognitive functions, and rule deduction. The VRCTI comprised 12 different tasks distributed in 8 sessions with different difficulty levels. The passive control group received usual care. Older adults were randomly assigned to either VR or control groups. An experimental pre-post design was used. Accuracy, error, and repetition rates were measured throughout each session. Intervention effects were analyzed using a generalized estimating equation model.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years
* Admitted as residents at the study-site institutions (long-term care facilities)
* Mini Mental Status Examination (MMSE) ≥ 13
* Able to communicate sufficiently

Exclusion Criteria:

* Open facial wounds
* Problems with a finger, hand, or wrist and/or major visual or auditory impairment, making it difficult to deliver training scheme
* Major neurological or psychiatric conditions that may affect cognition (e.g., stroke, dizziness, schizophrenia)
* Unstable medical conditions
* Were unable to comply with the intervention

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Cognitive Assessment Screening Instrument (CASI) | Change is being assessed. Change in Cognitive Assessment Screening Instrument (CASI) from baseline to immediately after the intervention.
  The CASI evaluates global cognitive function using 9 cognitive domains: long-term memory, short-term memory, attention, mental manipulation, orientation, abstraction and judgment, language abilities, visual construction, and list-generating fluency. Typical administration time is about 20 minutes. The total score ranges from 0 to 100. A greater score demonstrates better global cognitive function.
Mini-Mental State Examination (MMSE) | Change is being assessed. Change in Mini-Mental State Examination (MMSE) from baseline to immediately after the intervention.
  General cognitive functioning was assessed with the Chinese version of the MMSE, which is a cognitive screening tool used to evaluate cognitive decline, screen for cognitive impairment, to evaluate the severity of the impairment, and to monitor cognitive change over time. The higher score indicates the better cognitive function.
Clock Drawing Test-Drawing Part, (CDT-D) | Change is being assessed. Change in Clock Drawing Test-Drawing Part, (CDT-D) from baseline to immediately after the intervention.
  The CDT-D has been widely used as a neuropsychological screening test in the detection of cognitive impairment in populations. The lower the patients' clock scores the more likely were patients to be classified as impaired in elderly outpatients.
World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF) | Change is being assessed. Change in World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF) from baseline to immediately after the intervention.
  The WHOQOL-BREF contains 28 items classified into the same 4 domains related to quality of life (physical health, psychological, social relationships and environment). All items were rated on a 5-point scale with a higher score indicating a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chi Hsu, Ph.D, Principal Investigator — I-Shou University
Locations (1):
- I-Shou University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data presented in this study are available on request from the researcher. The data are not publicly available due to privacy and ethical restrictions.